CLINICAL TRIAL: NCT06456476
Title: Study Of Patients With Obstructive Jaundice In Sohag University Hospital
Brief Title: Patients With Obstructive Jaundice In Sohag University Hospital
Acronym: Jaundice
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Al Shaimaa Ibrahim Hamdy, principal investigator, Sohag University
Other Study IDs: Soh-Med-24-04-03MS
Record Dates: First submitted 2024-05-27; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Jaundice
MeSH Terms: conditions — Jaundice, Obstructive | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patints with obstructive jaundicep: The patients, clinically diagnosed as suffering from obstructive jaundice and referred to the Department of Internal Medicine for further evaluation.
  Interventions: Diagnostic Test: ERCP

INTERVENTIONS:
Diagnostic Test: ERCP — ERCP used only if needed in some patients

SUMMARY:
Study of patients with obstructive jaundice in Sohag university hospital study the clinical, laboratory and imaging charachteristics in patients with obstructive jaundice admitted to sohag university hospital, and to study the available therapeutic options which meight improve patient's quality of life and increase survival rates.

DETAILED DESCRIPTION:
Jaundice is always a pathological sign on most occasions, so that it should never be ignored. It includes 3 types: haemolytic, hepatocellular and cholestatic (obstructive).

Cholestatic jaundice can be classified into two broad categories: intrahepatic and extrahepatic; Intrahepatic cholestatic jaundice is due to impaired hepatobiliary production and excretion of bile causing bile components to enter the circulation. The concentration of conjugated bilirubin in serum is elevated in cholestatic jaundice. Intrahepatic cholestasis may be due to primary biliary cirrhosis, hepatocellular disease such as acute viral hepatitis infection, drug-induced liver injury ,Dubin-Johnson syndrome, Rotor syndrome, or cholestatic disease of pregnancy. Wilson's disease may also lead to intrahepatic cholestasis due to copper deposition into liver parenchyma, with further hepatocellular dysfunction, and jaundice.1 Extrahepatic cholestasis may be the result of benign causes including choledocholithiasis (is the most frequent cause), primary sclerosing cholangitis, Mirrizi syndrome, postoperative billiary stricture, post inflammatory stricture, pancreatitis, choledochal cyst, pyogenic cholangitis, parasitic diseases, duodenal diverticulosis and AIDS cholangiopathy.2 While malignant causes include cancer head of pancreas, carcinoma of the gall bladder cholangiocarcinoma, carcinoma of the duodenum, ampullary tumors, hepatocellular carcinoma, lymphoma and metastatic tumors.3 Today's obstructive jaundice is more of a medical entity since gastroenterologists, rather than surgeons, handle the majority of obstructive jaundice cases with ERCP or stenting.4 Obstructive jaundice patients typically complain of jaundice, yellowish discoloration of skin and eyes, pruritus, clay colored stool, dark-colored urine and aneroxia.5 Jaundice in choledocholithiasis is intermittent and associated with pain.6-7 Malignant jaundice commonly presents with persistent and progressive painless jaundice, often accompanied by weight loss, anemia, and abdominal mass.6-8 Patients with obstructive jaundice are susceptible to developing deficiencies in nutrition, infectious complications , acute renal failure, and compromised cardiovascular function. Other adverse events , like endotoxemia, hypovolemia, and coagulopathy, can be subtle and dramatically raise mortality and morbidity.9 A combination of many approaches, such as the patient's history, physical examination, biochemical tests, and imaging are needed. Abdominal ultrasonography, the first-line imaging modality used for the diagnosis of obstructive jaundice because it is noninvasive, fast and widely accessible.10 However, it is necessary to combine ultrasonography with other imaging techniques such as; computed tomography (CT), endoscopic ultrasonography (EUS) or magnetic resonance cholangiography (MRCP) to establish local and distant complications and make a choice of the right therapeutic approach.11 also liver biopsy, as well as observation of patient's course, can lead to an accurate diagnosis.

Early and precise detection of etiology of obstructive jaundice can help to manage such patients and thus will enhance the patient's quality of life and increase the survival rate of patients with malignant pathology.12

ELIGIBILITY:
Inclusion Criteria:

* The patients, clinically diagnosed as suffering from obstructive jaundice and referred to the Department of Internal Medicine for further evaluation.

Exclusion Criteria:

* Exclusion criteria were patients below 18 years of age; and patients with jaundice due to causes other than obstructive pathology like hemolytic or hepatocellular jaundice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients, clinically diagnosed as suffering from obstructive jaundice and referred to the Department of Internal Medicine for further evaluation.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Study Of Patients With Obstructive Jaundice In Sohag University Hospital | 6 months
  rate of patients with obstructive jaundice admitted in sohag university hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] deLemos AS, Ghabril M, Rockey DC, Gu J, Barnhart HX, Fontana RJ, Kleiner DE, Bonkovsky HL; Drug-Induced Liver Injury Network (DILIN). Amoxicillin-Clavulanate-Induced Liver Injury. Dig Dis Sci. 2016 Aug;61(8):2406-2416. doi: 10.1007/s10620-016-4121-6. Epub 2016 Mar 22. PMID 27003146
- [Background] Roche SP, Kobos R. Jaundice in the adult patient. Am Fam Physician. 2004 Jan 15;69(2):299-304. PMID 14765767
- [Background] Moghimi M, Marashi SA, Salehian MT, Sheikhvatan M. Obstructive jaundice in Iran: factors affecting early outcome. Hepatobiliary Pancreat Dis Int. 2008 Oct;7(5):515-9. PMID 18842499
- [Background] Qin LX, Tang ZY. Hepatocellular carcinoma with obstructive jaundice: diagnosis, treatment and prognosis. World J Gastroenterol. 2003 Mar;9(3):385-91. doi: 10.3748/wjg.v9.i3.385. PMID 12632482